CLINICAL TRIAL: NCT06738641
Title: The Effects of a Digital Customized Healthy Habit Software (Pro2col Health) on Health-Related Habits, Healthspan, and Biological Age
Brief Title: Effects of Pro2col Application on Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science & Performance Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P083124
Record Dates: First submitted 2024-12-10; First posted 2024-12-17 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Health Behavior; Nutrition, Healthy; Activity, Motor
MeSH Terms: conditions — Health Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled parallel study with pre- and post-measures
Masking Description: This is an open trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pro2col (Experimental): The experimental group will be enrolled in the Prime Health Technologies software (Pro2col), which provides a digital diagnostic score to calculate healthspan and biological age, along with AI and group community-based coaching dynamics. Subjects will be assigned a 6 week progressive protocol targeting improvements in daily activity levels, nutritional awareness, and overall lifestyle risk factors.
  Interventions: Behavioral: Pro2col Health
- Control (Active Comparator): The control group will receive subject-facing materials depicting current general activity recommendations as published by the American Heart Association (AHA) and current dietary guidelines provided by the United States Department of Agriculture (USDA).
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Pro2col Health — The Pro2col Health application is a smartphone application that provides users with health behavior guidance, personalized feedback, and assessments designed to estimate their current healthspan and biological age.
  Arms: Pro2col
Behavioral: Control — The control group will receive subject-facing materials depicting current general activity recommendations as published by the American Heart Association (AHA) and current dietary guidelines provided by the United States Department of Agriculture (USDA).
  Arms: Control

SUMMARY:
The purpose of this study is to test the effectiveness of a novel smartphone application (Pro2col Health) in regard to multiple health outcomes and health behaviors in healthy middle-aged adults.

DETAILED DESCRIPTION:
This is a non-blinded randomized controlled pilot trial conducted over up to 8 weeks. Week 0 will involve baseline measurements and enrollment, Weeks 1-6 constitute the intervention, and Week 7 to 8 is reserved for post-testing. The study will enroll up to 200 participants, with a minimum of 50 participants who meet the inclusion criteria, and a minimum target of 20 participants completing the study in each group (experimental and control).

Following baseline testing and enrollment in the study, participants will be randomly assigned to either the control (CON) or experimental (PRO) group. The control group will receive subject-facing materials depicting current general activity recommendations as published by the American Heart Association (AHA) and current dietary guidelines provided by the United States Department of Agriculture (USDA). The experimental group will be enrolled in the Prime Health Technologies software (Pro2col), which provides a digital diagnostic score to calculate healthspan and biological age, along with AI and group community-based coaching dynamics. Subjects will be assigned a 6 week progressive protocol targeting improvements in daily activity levels, nutritional awareness, and overall lifestyle risk factors. Both groups will then be monitored by study staff throughout the duration of the intervention period with post-testing taking place following the last week of the experiment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 21-60 years.
* A BMI categorized as overweight (≥ 25) but not stage II obesity (≤ 35)
* Daily steps < 5,000.
* Ownership of a smartphone device with either the Apple Health or Google Fit application.
* Willingness to carry their phone in their pocket or on their person at all times to track steps during study.
* Willing to download the Pro2col application and connect it with either the Apple Health or Google Fit application.
* Willingness to complete physical tasks including a timed one-mile walk/run, regular or modified push-ups to exhaustion, and chair get-ups to exhaustion.
* For the experimental group, subjects must be willing to follow the application protocol.
* Able to read, understand, sign and date the informed consent document (English only)
* Able and willing to comply with the scheduled visit(s) and study requirements.

Exclusion Criteria:

* Currently taking (within the past 30 days) ergogenic dietary supplements including, creatine, protein, amino acids, or stimulants other than caffeine (yohimbe, ephedrine, etc.) Currently taking performance enhancing drugs (testosterone or other anabolic-androgenic steroids), human growth hormone, insulin, etc.
* History or current malignancy
* Receiving chemotherapy agents or radiation treatments
* Musculoskeletal disease (muscular dystrophy, arthritis, etc.)
* Recent (<3-months) musculoskeletal injuries
* BMI < 25 or > 35 kg/m2
* Diagnosis of a terminal illness
* Use of prescription medications that influence body composition (i.e., prescription hormone therapies, etc.)
* History of alcohol abuse
* History or current drug abuse
* History or current diagnosis of depression.
* History or current diagnosis of suicidal thoughts/ideation.
* A score of ≥ 10 arbitrary units on the PHQ-9 during baseline testing.
* History or current cigarette smoke (including vaping) within the past 14 days from the screening visit
* Insulin-dependent diabetes and/or metformin use
* Chronic kidney or liver disease
* Has significant concurrent illnesses (controlled or uncontrolled), such as diabetes, lupus, epilepsy, or cardiac disorders, hepatitis B/C, HIV, serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in the past two years, or other, which in the opinion of the investigator, such conditions might be aggravated as a result of treatment
* The investigator feels that for any reason the subject is not eligible to participate in the study
* History of uncontrolled cardiovascular disease (i.e., myocardial infarction, hypertension, hypercholesterolemia, peripheral vascular disease, other)
* Developmental disability or cognitive impairment that would preclude adequate comprehension of the informed consent form and/or ability to follow study subject requirement and/or record the necessary study measurements
* A family member of the investigator or an employee of the investigator
* Participation in any other investigational study within 30 days prior to consent.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-10-06 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Biological Age | 6-weeks
  Assessed via a proprietary algorithm sourced within the application.
Muscle Strength-Endurance | 6-weeks
  Assessed by performance measures including push-ups to exhaustion, and chair get-ups to exhaustion.
Body Composition | 6-weeks
  Assessed via a previously validated digital scale.
Blood Pressure | 6-weeks
  Assessed via an electronic blood pressure cuff.
Daily Steps | 6-weeks
  Collected via the Apple Health or Google Fit application on the subject's pre-existing personal device.
Physical Endurance | 6-weeks
  Assessed via a one mile walk time.

SECONDARY OUTCOMES:
Depression | 6-weeks
  Assessed by the previously validated Patient Health Questionnaire 9 (PHQ-9) subjective questionnaire. Scores from each question are summed for a total of 0 to 27 points, with higher scores representing more symptoms of depression.
Quality of Life (SF-36 Survey) | 6-weeks
  Assessed by the previously validated Short Form 36 (SF-36) subjective questionnaire. This questionnaire houses 8 unique domains of quality of life measures, and each domain is scored from 0-100 based on subject responses (higher scores represent better quality of life). Scores from all 8 domains are then averaged to provide an aggregate score for the SF-36.

CONTACTS AND LOCATIONS:
Locations (1):
- Applied Science and Performance Institute, Tampa, Florida, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT06738641/Prot_SAP_000.pdf